CLINICAL TRIAL: NCT03167827
Title: Effects of Physical Training and Isoflavone Supplementation On Pelvic Floor Musculature in Women in the Postmenopausal Period: Controlled Randomized Clinical Trial
Brief Title: Effects of Physical Training and Isoflavone Supplementation On Pelvic Floor in Women in the Postmenopausal Period
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Natasha Morena Bazílio Silva, physiotherapist, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP UFU 52969515.1.0000.5152
Record Dates: First submitted 2017-05-17; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Pelvic Floor
Keywords: pelvic floor; climateric; exercise; Supplementation of Isoflavone
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Isoflavones

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider
Masking Description: Double Blind (Participant, Care Provider)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group isoflavone and exercise (Experimental): The isoflavone group received daily 100mg of isoflavones.
  Interventions: Other: Exercise; Other: isoflavone
- Group placebo and exercise (Placebo Comparator): The placebo group received 100mg containing starch of corn.
  Interventions: Other: Exercise; Other: placebo

INTERVENTIONS:
Other: Exercise — The training program consisted of aerobic and resisted combined physical exercises performed during 10 weeks, three times weekly with 45 minutes sessions: 5 minutes of warm-up on treadmill, 20 minutes of aerobic exercises and 20 minutes of resistance exercises.
Other: isoflavone — Daily supplementation in 1 capsule per day of 100mg of isoflavones (containing 3.3% genistein, 93.5% dadzein and 3.2% glycitein).
  Arms: Group isoflavone and exercise
Other: placebo — Daily supplementation in 1 capsule per day containing starch of corn.
  Arms: Group placebo and exercise

SUMMARY:
This study evaluates the effect of Physical Training and Supplementation of Isoflavone About Pelvic Floor Musculature in Women in the Postmenopausal period, and it has two groups the intervetion.

DETAILED DESCRIPTION:
The practice of physical exercise and isoflavone supplementation are ways of treating symptoms of climacteric, there is a lack of evidence as to whether these therapeutics when associated are useful for improving the strength, function, contraction pressure, electrical activity of the pelvic floor musculature of women in the Postmenopausal period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal woman
* to be able to practice exercises on treadmill and weight exercises
* without physical complications that prevent the execution of physical exercises
* have no history of cardiovascular disease, diabetes, renal pathologies or hypertension
* Present ability to contract the pelvic floor muscles

Exclusion Criteria:

* Smokers
* Use hormone therapy or isoflavone
* Use drugs that interfere with lipid and antihypertensive metabolism
* Presence of cognitive impairment or neurological condition that could affect muscle activation
* Present urinary tract infection at the time of data collection
* Training pelvic floor muscle

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The change vaginal squeeze pressure | before and after the intervetion ( 10 weeks)
  The vaginal squeeze pressure was measured through Perineometer.To obtain the measurements, the subjects remained positioning and vaginal sensor was introduced into the vaginal cavity. The women were oriented and motivated verbally to perform three voluntary maximal contractions sustained for five seconds and one minute interval between them. Outcome Measure of the vaginal squeeze pressure is cmH20 or Pascal.
The change Muscle function | before and after the intervetion (10 weeks)
  "PFM" evaluation was performed by vaginal palpation .During vaginal palpation the physiotherapist introduced the index and middle fingers about 4cm inside the vagina, and requested to hold the maximum contraction of the "PFM". Muscle function was classified by the Oxford Scale Modified that five grades of the force.
The change electromyography pelvic floor | before and after the intervetion (10 weeks)
  "PFM" electromyographic activity was collected during the resting to normalize the EMG data. No instruction regarding "PFM" contraction was given during the resting of the eight seconds. After, the volunteers were instructed to perform a maximal voluntary "PFM" contraction with the instruction to move "inward and upward" with the greatest possible force and to hold the contraction for five seconds. The women were oriented and motivated verbally to perform three voluntary maximal contractions sustained for five seconds and one minute interval between them.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arab AM, Behbahani RB, Lorestani L, Azari A. Correlation of digital palpation and transabdominal ultrasound for assessment of pelvic floor muscle contraction. J Man Manip Ther. 2009;17(3):e75-9. doi: 10.1179/jmt.2009.17.3.75E. PMID 20046616
- [Result] Pereira VS, Hirakawa HS, Oliveira AB, Driusso P. Relationship among vaginal palpation, vaginal squeeze pressure, electromyographic and ultrasonographic variables of female pelvic floor muscles. Braz J Phys Ther. 2014 Sep-Oct;18(5):428-34. doi: 10.1590/bjpt-rbf.2014.0038. Epub 2014 Oct 10. PMID 25372005
- [Result] Bo K, Finckenhagen HB. Vaginal palpation of pelvic floor muscle strength: inter-test reproducibility and comparison between palpation and vaginal squeeze pressure. Acta Obstet Gynecol Scand. 2001 Oct;80(10):883-7. doi: 10.1034/j.1600-0412.2001.801003.x. PMID 11580731